CLINICAL TRIAL: NCT04548466
Title: Effect of Positive Expiratory Pressure on the Management of Chest Trauma: a Randomized Controlled Trial
Brief Title: Effect of Positive Expiratory Pressure on the Management of Chest Trauma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital de Granollers (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CT-positive expiratory
Record Dates: First submitted 2020-09-07; First posted 2020-09-14 (Actual); Last update posted 2020-09-14 (Actual); Status verified 2020-09

CONDITIONS: Thoracic Fracture

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CONTROL group (No Intervention): Chest physiotherapy depending on the location of the ribs fractures techniques are performed: 1. Postural control techniques; 2. Airways clearance techniques; 3. Breathing exercise (diaphragmatic breathing). 4. Early mobilization.
- PEP group (Experimental): Chest physiotherapy depending on the location of the ribs fractures techniques are performed: 1. Postural control techniques; 2. Airways clearance techniques; 3. Breathing exercise (diaphragmatic breathing). 4. Early mobilization. 5. Positive expiratory pressure breathing (PEP bottle)
  Interventions: Device: PEP bottle

INTERVENTIONS:
Device: PEP bottle
  Arms: PEP group

SUMMARY:
Chest trauma (CT) are a common problem in our environment caused mainly by traffic accidents and causal and domestic accidents among the elderly population. CTs, in some situations, can lead to sequelae such as fibrothorax secondary to hemothorax and / or empyema and residual chronic pain. Clinical regulations and guidelines recommend a guideline for chest physiotherapy (CP) for all patients with rib fractures, but there is little scientific evidence. It would be interesting to establish CP treatment protocols and describe the most appropriate techniques according to the type and stages of thoracic trauma consolidation.

Objective: To evaluate the effect of Positive Expiratory Pressure (PEP) breathing added to conventional CP in terms of aid secretion clearance, pain control, pleuropulmonary radiological abnormalities, restoration of lung function, and admission days in the immediate phase of the CT.

DETAILED DESCRIPTION:
After acceptance to participate in the study, patients will be computerized randomized into 2 groups:

* PEP group: positive expiratory pressure breathing.
* CONTROL group: conventional CP treatment without positive pressure brething. The period between day 0 and 20 days post-trauma is considered an immediate phase of CT.

Once admitted, an initial evaluation by the doctor will be performed, and pleuro-pulmonary complications, the presence of respiratory failure, and pain control will be evaluated. The chest physiotherapist will perform a clinical and secretion assessment using the Seva test and a dynamic costal examination. The medical treatment of pain control will begin, and the treatment of CP will begin, where it will be randomized in 2 groups: 1- PEP group: positive expiratory pressure breathing with the help of a PEP bottle device. 2-CONTROL group: conventional CP treatment without positive pressure breathing will be daily FR sessions, on weekdays. Upon admission, hospital discharge and post-discharge, radiological checks (simple radiography) will be performed and forced vital capacity will be measured with forced spirometry.

ELIGIBILITY:
Inclusion Criteria:

* Chest trauma with three or more rib fractures with or without hemopneumothorax
* Failure to meet any exclusion criteria

Exclusion Criteria:

* Non-cooperative patients for not understanding chest physiotherapy techniques.
* Presence of respiratory failure on admission: PaO2 <60mmHg i / or PaCO2> 50mmHg.
* Medical indication for mechanical ventilation or non-invasive ventilatory support.
* Presence of undrained pneumothorax.
* Complications that limit early mobility.

Ages: 18 Years to 88 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2015-10 (Actual); Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Aid secretion clearance | 1 month
  To determine if PEP bottle improves the secretion clearance

SECONDARY OUTCOMES:
Resolution of pleural lesions | 1 month
  To analysed if PEP bottle allows faster resolution of pleural lesions
Improve lung function | 1 month
  To determine if PEP bottle improves lung function tests
Reduce hospital stay | 1 month
  To assess if PEP bottle decreased hospital stay

CONTACTS AND LOCATIONS:
Overall Officials: Gemma Molist, Study Chair — Hospital de Granollers
Locations (1):
- Inmaculada Castillo, Seva, Barcelona, Spain

REFERENCES:
- [Background] Dogrul BN, Kiliccalan I, Asci ES, Peker SC. Blunt trauma related chest wall and pulmonary injuries: An overview. Chin J Traumatol. 2020 Jun;23(3):125-138. doi: 10.1016/j.cjtee.2020.04.003. Epub 2020 Apr 20. PMID 32417043
- [Background] Liebsch C, Seiffert T, Vlcek M, Beer M, Huber-Lang M, Wilke HJ. Patterns of serial rib fractures after blunt chest trauma: An analysis of 380 cases. PLoS One. 2019 Dec 19;14(12):e0224105. doi: 10.1371/journal.pone.0224105. eCollection 2019. PMID 31856165
- [Background] Ingoe HM, Coleman E, Eardley W, Rangan A, Hewitt C, McDaid C. Systematic review of systematic reviews for effectiveness of internal fixation for flail chest and rib fractures in adults. BMJ Open. 2019 Apr 1;9(4):e023444. doi: 10.1136/bmjopen-2018-023444. PMID 30940753
- [Background] Witt CE, Bulger EM. Comprehensive approach to the management of the patient with multiple rib fractures: a review and introduction of a bundled rib fracture management protocol. Trauma Surg Acute Care Open. 2017 Jan 5;2(1):e000064. doi: 10.1136/tsaco-2016-000064. eCollection 2017. PMID 29766081
- [Background] Gunduz M, Unlugenc H, Ozalevli M, Inanoglu K, Akman H. A comparative study of continuous positive airway pressure (CPAP) and intermittent positive pressure ventilation (IPPV) in patients with flail chest. Emerg Med J. 2005 May;22(5):325-9. doi: 10.1136/emj.2004.019786. PMID 15843697
- [Background] Sehlin M, Ohberg F, Johansson G, Winso O. Physiological responses to positive expiratory pressure breathing: a comparison of the PEP bottle and the PEP mask. Respir Care. 2007 Aug;52(8):1000-5. PMID 17650355